CLINICAL TRIAL: NCT00269061
Title: An Exploratory MRI Study in Type 2 Diabetic Subjects: A Randomized, Double-Blinded, Placebo-Controlled Trial to Evaluate the Measurement of Fluid Volumes by MRI in the Lower Extremities of Subjects Receiving Pioglitazone
Brief Title: Study In Patients With Type 2 Diabetes Who Are Taking Metformin And Sulfonylurea, Metformin And Insulin, Or Insulin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADG104148
Record Dates: First submitted 2005-12-22; First posted 2005-12-23 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: Non-Insulin-Dependent Diabetes Mellitus
Keywords: pioglitazone; diabetes; fluid
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Pioglitazone

INTERVENTIONS:
Drug: pioglitazone

SUMMARY:
This study will use Magnetic Resonance Imaging (MRI) techniques to evaluate changes in fluid volume in the lower legs of diabetic patients who add either pioglitazone or placebo to their current diabetic regimen.

ELIGIBILITY:
Inclusion criteria:

* Must have been diagnosed with Type 2 diabetes at least three months prior to screening.
* Must be taking either metformin and a sulfonylurea, metformin and insulin, or insulin only, and doses of these medications must have been stable for at least three months.
* Must have a Body Mass Index (BMI) of between 24 and 35.
* If female, the subject must be post-menopausal.
* HbA1c levels must be between 7% and 10%.
* Subjects must be eligible for MRI scanning (ie, no metal implants, pacemaker, etc).

Exclusion criteria:

* Suffer from claustrophobia.
* Use of tobacco, nicotine, or illegal drugs of abuse.
* Use of caffeine within two days prior to each study visit.
* HIV, hepatitis, edema, untreated blood pressure problems, heart, lung, nervous system or kidney disease, history of blood clots in the legs, diabetic neuropathy, or untreated thyroid disease.
* Use of drugs or medications that affect the levels of fluid in the body, such as diuretics.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32
Dates: Start 2006-01

PRIMARY OUTCOMES:
Changes in interstitial fluid volume in the lower extremities as measured by MRI.

SECONDARY OUTCOMES:
Assessments of other indicators of fluid volume changes, including labwork evaluation, fluid compartment volume measurement, direct measurement of the calf.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Belmont, Massachusetts, United States